CLINICAL TRIAL: NCT03016169
Title: Trifecta™ GT (Glide Technology) Post Market Clinical Follow-up (PMCF)
Brief Title: Trifecta™ GT Post Market Clinical Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10120
Record Dates: First submitted 2016-12-21; First posted 2017-01-10 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Disease; Aortic Valve Disorder
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Other): All subjects will receive the Trifecta GT valve
  Interventions: Device: Trifecta GT (Glide Technology) Valve

INTERVENTIONS:
Device: Trifecta GT (Glide Technology) Valve — Surgical aortic valve replacement with Trifecta GT Valve.

SUMMARY:
The objective of this study is to evaluate the safety and performance of the Trifecta™ GT (Glide Technology) valve through 5 year follow-up in a prospective, multi-center, real-world setting. This study is intended to satisfy post-market clinical follow-up requirements of CE Mark in Europe.

DETAILED DESCRIPTION:
The study is a prospective multi-center evaluation of approximately 350 subjects implanted with a St. Jude Medical (SJM) Trifecta™ GT valve. It will be conducted in approximately 35 sites worldwide.

Subjects will be followed for 5 years. The total duration of the study is expected to be 6 years, assuming all subjects are enrolled within 1 year of study initiation. To ensure enrollment balance across sites, no individual site can enroll more than 10% of the sample size (n=35 subjects) without prior approval from the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a candidate for surgical aortic valve replacement per current guidelines and is intended to be implanted with a St. Jude Medical Trifecta GT valve.
2. Subject is of legal age in the country where the subject is enrolled.
3. Subject must be willing and able to provide written informed consent to participate in this study.
4. Subject must be willing and able to comply with all follow-up requirements.

Exclusion Criteria:

1. Subject undergoes a concomitant procedure of mitral or tricuspid valve replacement at the time of the Trifecta GT valve implantation surgery.
2. Subject has contraindication for cardiac surgery.
3. Subject is pregnant. Pregnancy will be assessed by the subject informing the physicians.
4. Subject has active endocarditis (subjects who have previously experienced endocarditis must have two documented negative blood culture results while off antibiotic therapy prior to the valve implantation surgery).
5. Subject has had a stroke or transient ischemic attack within 6 months prior to the planned valve implantation surgery.
6. Subject is undergoing renal dialysis.
7. Subject has a history of active drug addiction, active alcohol abuse, or psychiatric hospital admission for psychosis within the prior 2 years.
8. Subject has a documented thrombus in the left atrium or left ventricle at the time of the valve implantation surgery.
9. Subject has a left ventricular ejection fraction < 30%.
10. Subject previously enrolled in the Trifecta GT PMCF study and withdrawn (a subject cannot be enrolled twice in this study).
11. Preoperative evaluation indicates other significant cardiovascular abnormalities such as aortic dissection or ventricular aneurysm.
12. Subject has a life expectancy less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, Study Director — Abbott Structural Heart
Locations (27):
- United States (5):
  - Mayo Clinic, Rochester, Minnesota
  - Mission Health & Hospitals, Asheville, North Carolina
  - Main Line Health Center/Lankenau Hospital, Wynnewood, Pennsylvania
  - Centennial Medical Center, Nashville, Tennessee
  - CHI St. Luke's Health Baylor College of Medicine, Houston, Texas
- Cliniques Universitaires Saint Luc, Brussels, Brussels Capital, Belgium
- Canada (3):
  - Saint John Regional Hospital - New Brunswick Heart Centre, Saint John, New Brunswick
  - Toronto General Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
- Tartu University Hospital, Tartu, Estonia
- CHRU Hopital de Pontchaillou, Rennes, Brittany Region, France
- Germany (6):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim, Hesse
  - Krankenhaus der Barmherzigen Brüder, Trier, Rhineland-Palatinate
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - Universitätsklinikum Jena, Jena, Thuringia
  - Deutsches Herzzentrum Berlin, Berlin
  - Asklepios Klinik Harburg, Hamburg
- Italy (3):
  - Ospedale Niguarda Ca'Granda, Milan, Lombardy
  - Az. Osp Universitaria Careggi, Florence, Tuscany
  - Ospedale dell'Angelo, Mestre, Veneto
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands
- Centralny Szpital Kliniczny MSW w Warszawie, Warsaw, Masovian Voivodeship, Poland
- Hospital de São João, Porto, Portugal
- Spain (2):
  - Hospital Universitario del Vinalopó, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Island
- United Kingdom (2):
  - Plymouth Hospitals NHS Trust - Derriford Hospital, Plymouth, South West England
  - St. Bartholomew's Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 358 subjects were enrolled across 27 investigational sites in 12 North American and European countries. The Trifecta GT PMCF study is a single-arm, prospective, multi-center clinical investigation designed to evaluate the five-year safety and performance of the Trifecta GT valve in patients indicated for aortic valve replacement.
Period: Overall Study
Arm/Group | Treatment
Started | 358
Completed | 269
Not Completed | 89
Not completed — Lost to Follow-up | 4
Not completed — Death | 54
Not completed — Device Explant | 11
Not completed — Withdrawal by Subject | 19
Not completed — Other Reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140
  Male | 218
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hypertension [Count of Participants; unit: Participants] | 291

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Surgical Valve Replacement or Transcatheter Valve-in-Valve Implantation
Description: Estimated percentage of participants free from undergoing an additional aortic valve replacement within 5 years, using a Kaplan-Meier estimate.
Time Frame: 5 years post implant
Population: Analysis population includes participants implanted with the Trifecta™ valve in the study on 10 March 2017 and continued through 05 February 2018.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 358
percentage of participants | 95.8 [92.8 to 97.6]

2. Other Pre Specified Outcome: Freedom From All-cause Mortality
Description: Estimated percentage of participants surviving at 5 years, using a Kaplan-Meier estimate.
Time Frame: 5 years post implant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 358
percentage of participants | 84.5 [80.2 to 88.0]

3. Other Pre Specified Outcome: Freedom From Valve Related Mortality
Description: Estimated percentage of participants remaining free from a valve-related death at 5 years, using a Kaplan-Meier estimate. The estimate includes subjects alive at 5 years and subjects who died for reasons unrelated to the valve at 5 years.
Time Frame: 5 years post implant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 358
percentage of participants | 95.4 [92.3 to 97.2]

4. Other Pre Specified Outcome: Freedom From Structural Valve Deterioration
Description: Estimated percentage of participants free from structural valve deterioration at 5 years, as using a Kaplan-Meier estimate. Structural valve deterioration is any change in function of the valve resulting in an intrinsic abnormality of the valve that causes stenosis or regurgitation.
Time Frame: 5 years post implant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 358
percentage of participants | 96.2 [93.3 to 97.9]

5. Other Pre Specified Outcome: Freedom From Surgical Valve Replacement or Transcatheter Valve Implantation Due to Structural Valve Deterioration
Description: Estimated percentage of participants who do not require surgery due to structural valve deterioration, using a Kaplan-Meier estimate.
Time Frame: 5 years post implant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 358
percentage of participants | 98.2 [95.8 to 99.3]

6. Other Pre Specified Outcome: Valve Hemodynamic Performance for Left Ventricular Ejection Fraction (LVEF) at Six Months
Description: LVEF is a measurement of the percentage of blood leaving the heart each time it contracts.
Time Frame: 6 Months
Population: Analysis population includes all study participants with an LVEF assessment at 6 months.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Treatment
Number analyzed (Participants) | 234
percentage | 60.4 (7.5)

7. Other Pre Specified Outcome: Valve Hemodynamic Performance for Effective Orifice Area (EOA) at Six Months
Description: EOA measures the functional valve opening for blood flow through the valve.
Time Frame: 6 Months
Population: Analysis population includes all study participants with an EOA assessment at 6 months.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Treatment
Number analyzed (Participants) | 285
cm^2 | 2.0 (0.6)

8. Other Pre Specified Outcome: Valve Hemodynamic Performance for Indexed Effective Orifice Area (iEOA) at Six Months
Description: iEOA adjusts the EOA measurement to the patient's body size.
Time Frame: 6 Months
Population: Analysis population includes all study participants with an iEOA assessment at 6 months.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Treatment
Number analyzed (Participants) | 265
cm^2/m^2 | 1.0 (0.3)

9. Other Pre Specified Outcome: Valve Hemodynamic Performance for Mean Gradient at Six Months
Description: Mean Gradient measures the average pressure difference across the valve during blood flow.
Time Frame: 6 Months
Population: Analysis population includes all study participants with a mean gradient assessment at 6 months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment
Number analyzed (Participants) | 303
mmHg | 8.7 (3.3)

10. Other Pre Specified Outcome: Valve Hemodynamic Performance for Peak Gradient at Six Months
Description: Peak Gradient measures the maximum pressure difference across the valve during blood flow.
Time Frame: 6 Months
Population: Analysis population includes all study participants with a peak gradient assessment at 6 months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment
Number analyzed (Participants) | 302
mmHg | 16.6 (6.3)

ADVERSE EVENTS:
Time Frame: 5 Years
Description: All AEs reported in the Trifecta GT PMCF study.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 54/358
Serious Adverse Events (participants affected / at risk) | 206/358
Other Adverse Events (participants affected / at risk) | 82/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=358)
MAJOR BLEEDING - MEDIASTINAL OR THORACIC BLEED (Blood and lymphatic system disorders) | 2
MAJOR BLEEDING - OTHER BLEEDING (Blood and lymphatic system disorders) | 2
OTHER CARDIOVASCULAR (Blood and lymphatic system disorders) | 12
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Blood and lymphatic system disorders) | 7
EMBOLISM (Cardiac disorders) | 1
ENDOCARDITIS (Cardiac disorders) | 8
MAJOR BLEEDING - MEDIASTINAL OR THORACIC BLEED (Cardiac disorders) | 3
NONSTRUCTURAL DYSFUNCTION (Cardiac disorders) | 2
OTHER CARDIOVASCULAR (Cardiac disorders) | 83
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Cardiac disorders) | 3
STRUCTURAL VALVE DETERIORATION (Cardiac disorders) | 8
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Ear and labyrinth disorders) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Endocrine disorders) | 1
OTHER NEUROVASCULAR (Eye disorders) | 2
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Eye disorders) | 4
MAJOR BLEEDING - GASTROINTESTINAL BLEED (Gastrointestinal disorders) | 4
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Gastrointestinal disorders) | 17
OTHER CARDIOVASCULAR (General disorders) | 3
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (General disorders) | 11
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Hepatobiliary disorders) | 7
ENDOCARDITIS (Infections and infestations) | 8
OTHER CARDIOVASCULAR (Infections and infestations) | 3
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Infections and infestations) | 36
MAJOR BLEEDING - MEDIASTINAL OR THORACIC BLEED (Injury, poisoning and procedural complications) | 2
MAJOR BLEEDING - OTHER BLEEDING (Injury, poisoning and procedural complications) | 4
OTHER CARDIOVASCULAR (Injury, poisoning and procedural complications) | 3
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Injury, poisoning and procedural complications) | 6
OTHER CARDIOVASCULAR (Metabolism and nutrition disorders) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Metabolism and nutrition disorders) | 9
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Musculoskeletal and connective tissue disorders) | 16
OTHER NEUROVASCULAR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26
EMBOLISM (Nervous system disorders) | 3
MAJOR BLEEDING - OTHER BLEEDING (Nervous system disorders) | 1
OTHER CARDIOVASCULAR (Nervous system disorders) | 2
OTHER NEUROVASCULAR (Nervous system disorders) | 20
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Nervous system disorders) | 5
OTHER NEUROVASCULAR (Psychiatric disorders) | 3
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Psychiatric disorders) | 4
MAJOR BLEEDING - UROLOGIC BLEEDING (Renal and urinary disorders) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Renal and urinary disorders) | 18
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Reproductive system and breast disorders) | 3
MAJOR BLEEDING - MEDIASTINAL OR THORACIC BLEED (Respiratory, thoracic and mediastinal disorders) | 1
OTHER CARDIOVASCULAR (Respiratory, thoracic and mediastinal disorders) | 9
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Respiratory, thoracic and mediastinal disorders) | 31
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Skin and subcutaneous tissue disorders) | 2
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Social circumstances) | 1
MAJOR BLEEDING - MEDIASTINAL OR THORACIC BLEED (Surgical and medical procedures) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Surgical and medical procedures) | 4
EMBOLISM (Vascular disorders) | 9
MAJOR BLEEDING - MEDIASTINAL OR THORACIC BLEED (Vascular disorders) | 4
MAJOR BLEEDING - OTHER BLEEDING (Vascular disorders) | 3
OTHER CARDIOVASCULAR (Vascular disorders) | 7
OTHER NEUROVASCULAR (Vascular disorders) | 4
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Vascular disorders) | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=358)
OTHER CARDIOVASCULAR (Blood and lymphatic system disorders) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Blood and lymphatic system disorders) | 3
NONSTRUCTURAL DYSFUNCTION (Cardiac disorders) | 5
OTHER CARDIOVASCULAR (Cardiac disorders) | 42
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Cardiac disorders) | 2
STRUCTURAL VALVE DETERIORATION (Cardiac disorders) | 4
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Eye disorders) | 1
MAJOR BLEEDING - GASTROINTESTINAL BLEED (Gastrointestinal disorders) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Gastrointestinal disorders) | 3
OTHER CARDIOVASCULAR (General disorders) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (General disorders) | 2
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Infections and infestations) | 2
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Metabolism and nutrition disorders) | 2
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Musculoskeletal and connective tissue disorders) | 1
EMBOLISM (Nervous system disorders) | 2
OTHER NEUROVASCULAR (Nervous system disorders) | 3
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Nervous system disorders) | 2
NONSTRUCTURAL DYSFUNCTION (Product Issues) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Product Issues) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Psychiatric disorders) | 2
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Renal and urinary disorders) | 2
MAJOR BLEEDING - OTHER BLEEDING (Respiratory, thoracic and mediastinal disorders) | 1
OTHER CARDIOVASCULAR (Respiratory, thoracic and mediastinal disorders) | 1
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Respiratory, thoracic and mediastinal disorders) | 8
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Skin and subcutaneous tissue disorders) | 3
OTHER CARDIOVASCULAR (Vascular disorders) | 8
OTHER NON-CARDIOVASCULAR/NON-NEUROVASCULAR (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish study results until publication of results of multi center study or 2 years after study completion, whichever is sooner. PI allows Sponsor to review any proposed publication at least 40 days before forwarding it to any person that is not bound by confidentiality agreement between Sponsor and PI. Sponsor can request delay publication for no more than 120 days to allow Sponsor to file patent applications or take other measures to preserve or secure its Intellectual Property.

DOCUMENTS (2):
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT03016169/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT03016169/SAP_001.pdf